CLINICAL TRIAL: NCT00436969
Title: A Comparison of Orthovisc® to Corticosteroid Injection in Shoulder Osteoarthritis: Orthovisc Randomized Clinical Trial
Brief Title: ORTHOVISC Shoulder Osteoarthritis Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: DePuy Mitek (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06-OV-01
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Results first posted 2014-04-11 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2016-11

CONDITIONS: Glenohumeral Osteoarthritis
Keywords: Orthovisc; Osteoarthritis; Shoulder; Randomized
MeSH Terms: conditions — Osteoarthritis | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Subjects randomized to the control arm injection of prescribed anesthetic and corticosteroid, shall receive an equivalent volume (8 mL's).
  Interventions: Drug: Control
- Investigational (Experimental): Subjects randomized to the active treatment in this study will receive a one-time dose of 8 mL's of Orthovisc derived from non-animal source bacterial fermentation, S. Equi.
  Interventions: Device: Orthovisc

INTERVENTIONS:
Device: Orthovisc — Orthovisc injection
  Other Names: Hyaluronic acid
  Arms: Investigational
Drug: Control — Celestone (betamethasone sodium phosphate and acetate) - 2 mL
  Other Names: Corticosteroid
  Arms: Control

SUMMARY:
A comparison of Orthovisc to corticosteroid injections in the shoulder for pain due to osteoarthritis.

DETAILED DESCRIPTION:
This multicenter, prospective double-blinded, randomized trial will study two treatment groups. Subjects will be randomized to receive either Orthovisc or corticosteroids/anesthetic injection into the shoulder in a 2:1 schema. The trial will assess safety and efficacy of pain relief in the osteoarthritic shoulder.

ELIGIBILITY:
Inclusion Criteria:

* A candidate for unilateral treatment of osteoarthritis of the shoulder
* Have failed conservative treatment

Exclusion Criteria:

* Presence of full thickness Rotator Cuff tear and/or significantly compromised rotator cuff function
* No active instability or acute dislocation episodes within the previous 12 months
* Known allergy to hyaluronate preparations
* Pregnant or breast feeding
* Is receiving prescription pain medication for conditions unrelated to the index shoulder condition

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2006-12; Primary Completion 2010-02 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan B. McGlohorn, Study Director — DePuy Synthes Mitek and Biomaterials
Locations (13):
- United States (13):
  - CORE Orthopedics, Encinitas, California
  - Sierra Pacific Orthopaedic Center Medical Group, Fresno, California
  - UHZ Sports Medicine, Coral Gables, Florida
  - Andrews Research Institute, Gulf Breeze, Florida
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Massachusetts Merdical School - Worcester, Worcester, Massachusetts
  - Shores Rheumatology, Saint Clair Shores, Michigan
  - Insall Scott Kelly Institute, New York, New York
  - Tulsa Bone and Joint, Tulsa, Oklahoma
  - University Orthopedics Center, State College, Pennsylvania
  - The Methodist, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No
We will not submit the data to FDA, and as such will not be making IPD available.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between January 2007 and February 2010 at 13 sites based in the US.
Pre-assignment Details: Four subjects were randomized; however due to required imaging inclusion/exclusion criteria was not met. Hence, these 4 subjects were not treated.
Groups:
- Control: Each subject received a one-time injection containing 6 mL of anesthetic (Marcaine) and 2 mL of corticosteroid (Celestone).
- Investigational: Each subject received a one-time injection of 8 mL's of Orthovisc into the target shoulder.
Period: Overall Study
Arm/Group | Control | Investigational
Started | 88 | 186
Randomized But Not Treated | 1 | 3
Completed | 66 | 134
Not Completed | 22 | 52

BASELINE CHARACTERISTICS:
Population: The number of partipants analyzed were all 270 subjects that received treatment (87 control, 183 investigational).
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Investigational | Total
Number analyzed (Participants) | 87 | 183 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (9.84) | 58.6 (10.68) | 58.4 (10.40)
Age, Customized [Number; unit: participants]
  18 to 29 | 1 | 1 | 2
  30 and 39 years | 4 | 11 | 15
  40 to 49 years | 11 | 22 | 33
  50 to 59 years | 22 | 50 | 72
  60 to 69 years | 43 | 68 | 111
  70 to 79 years | 6 | 31 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 44 | 65
  Male | 66 | 139 | 205
Region of Enrollment [Number; unit: participants]
  United States | 87 | 183 | 270

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) Pain Score (Per Protocol)
Description: Scores are measured on a 100 mm Visual Analog Scale (VAS). The VAS scale ranges from 0 to 100 mm with the lower score indicating less pain and the higher score indicating greater pain.
Time Frame: 6 Months
Population: The Per Protocol analysis population was defined as all subjects that received treatment and completed 6 months of follow-up without a major protocol deviation.
Measure: Least Squares Mean (Standard Error); unit: mm on a 100 mm VAS scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 58 | 107
mm on a 100 mm VAS scale | 30.389 (3.035) | 28.917 (2.233)
Statistical Analysis 1: Comparison: Control vs Investigational; Anticipated VAS difference of 10 mm and SD of 25 mm indicated a sample size of 225 subjects in a 2:1 randomization would provide 80% power to detect a significant difference with a two-sided significance level of 5%. To account for a 15% dropout rate the sample size was increased to 270 subjects (180 Orthovisc, 90 control). The primary null hypothesis (Ho) no difference in VAS means at 6 months and the alternative hypothesis (Ha) was that Orthovisc (mean VAS) is superior to the control; Test type: Superiority or Other; p = 0.696, Mixed Models Repeated Measures ANCOVA — The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = -1.472, 95% CI 2-sided [-8.888 to 5.943]

2. Secondary Outcome: Percentage of Responders Using the Visual Analog Scale (VAS) Pain Score (Per Protocol)
Description: Scores are measured on a 100 mm Visual Analog Scale (VAS). The VAS scale ranges from 0 to 100 mm with the lower score indicating less pain and the higher score indicating greater pain.
  A responder was defined as a 20 mm or greater reduction in VAS pain score from baseline to 6 months.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Control | Investigational
Number analyzed (Participants) | 58 | 107
Percentage of Participants | 63.8 [50.1 to 76.0] | 63.6 [53.7 to 72.6]
Statistical Analysis 1: Comparison: Control vs Investigational; Asymptotic 95% confidence interval for the treatment group difference (Orthovisc - Control) in proportions of responders was calculated. The null hypothesis (Ho) is that the effect of the two treatment groups at 6 months is equal and the corresponding alternative hypothesis (Ha) is that the effect of the two treatment groups at 6 months is unequal; Test type: Superiority or Other; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-15.6 to 15.1]

3. Secondary Outcome: Percentage of Responders Using the Visual Analog Scale (VAS) Pain Score (As Treated)
Description: as for outcome 2
Time Frame: Baseline and 6 months
Population: The As Treated analysis population included all subjects that received treatment and had outcome data.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Control | Investigational
Number analyzed (Participants) | 67 | 136
Percentage of Participants | 59.7 [47.0 to 71.5] | 54.4 [45.7 to 63.0]
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -5.3, 95% CI 2-sided [-19.7 to 9.1]

4. Secondary Outcome: Visual Analog Scale (VAS) Pain Score Change From Baseline and 12 Weeks (Per Protocol)
Description: The difference in pain was calculated as visit score - baseline score. Scores are measured on a 100 mm visual analogy scale.
Time Frame: Baseline and 12 weeks
Population: The Per Protocol analysis population was defined as all subjects that received treatment and completed 6 months of follow-up without a major protocol deviation. Subjects were allowed to have missing interim visits (i.e. 12 weeks).
Measure: Least Squares Mean (Standard Error); unit: mm on a 100 mm VAS scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 49 | 91
mm on a 100 mm VAS scale | -23.624 (3.206) | -24.494 (2.356)
Statistical Analysis 1: Comparison: Control vs Investigational; The null hypothesis (Ho) is that the effect of the two treatment groups at 12 weeks is equal and the corresponding alternative hypothesis (Ha) is that the effect of the two treatment groups is unequal; Test type: Superiority or Other; p = 0.827, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = -0.870, 95% CI 2-sided [-8.698 to 6.957]

5. Secondary Outcome: Visual Analog Scale (VAS) Pain Score Change From Baseline and 12 Weeks (As Treated)
Description: Scores are measured on a 100 mm Visual Analog Scale (VAS). The VAS scale ranges from 0 to 100 mm with the lower score indicating less pain and the higher score indicating greater pain.
  The difference in pain was calculated as visit score - baseline score.
Time Frame: Baseline and 12 weeks
Population: The As Treated analysis population included all subjects that received treatment and had outcome data.
Measure: Least Squares Mean (Standard Error); unit: mm on a 100 mm VAS scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 65 | 135
mm on a 100 mm VAS scale | -16.882 (2.757) | -19.756 (1.909)
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.392, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = -2.875, 95% CI 2-sided [-9.472 to 3.723]

6. Secondary Outcome: American Shoulder and Elbow Surgeons Evaluation Form (ASES) Patient Score Change From Baseline and 12 Weeks (Per Protocol)
Description: The difference in American Shoulder and Elbow Surgeons Evaluation Form (ASES) Patient score calculated as visit score - baseline score.
  The ASES was designed to provide a standard method for evaluation of the shoulder through assessment of pain and activities of daily living (ie, function). The ASES is derived from an equation that incorporates a visual analog pain scale and functional ability questions. Both components have a maximum score of 50. Pain is calculated by subtracting the visual analog score from 10 and then multiplying by 5 for a total of 50 points. The function component is calculated by adding the points and multiplying by five thirds for a maximum of 50 points. The subscores for pain and function are then added for the total score. The maximum possible total score is 100, representing less pain and greater function.
Time Frame: Baseline and 12 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 41 | 75
units on a scale | 18.329 (2.578) | 17.397 (1.917)
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.772, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = -0.932, 95% CI 2-sided [-7.260 to 5.396]

7. Secondary Outcome: American Shoulder and Elbow Surgeons Evaluation Form (ASES) Patient Score Change From Baseline and 12 Weeks (As Treated)
Description: as for outcome 6
Time Frame: Baseline and 12 weeks
Population: The As Treated analysis population included all subjects that received treatment and had outcome data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 56 | 104
units on a scale | 12.960 (2.197) | 13.988 (1.605)
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.707, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = 1.028, 95% CI 2-sided [-4.338 to 6.393]

8. Secondary Outcome: American Shoulder and Elbow Surgeons Evaluation Form (ASES) Patient Score Change From Baseline and 6 Months (Per Protocol)
Description: as for outcome 6
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 50 | 84
units on a scale | 18.228 (2.438) | 17.408 (1.858)
Statistical Analysis 1: Comparison: Control vs Investigational; The null hypothesis (Ho) is that the effect of the two treatment groups at 6 months is equal and the corresponding alternative hypothesis (Ha) is that the effect of the two treatment groups is unequal; Test type: Superiority or Other; p = 0.790, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = -0.820, 95% CI 2-sided [-6.866 to 5.227]

9. Secondary Outcome: American Shoulder and Elbow Surgeons Evaluation Form (ASES) Patient Score Change From Baseline and 6 Months (As Treated)
Description: as for outcome 6
Time Frame: Baseline and 6 months
Population: The As Treated analysis population included all subjects that received treatment and had outcome data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 53 | 98
units on a scale | 14.272 (2.237) | 15.402 (1.636)
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.685, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = 1.130, 95% CI 2-sided [-4.341 to 6.001]

10. Secondary Outcome: Shoulder Pain and Disability Index (SPADI) Total Disability Score Change From Baseline and 12 Weeks (Per Protocol)
Description: The difference in Shoulder Pain and Disability Index (SPADI) Total Disability score calculated as visit score - baseline score.
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain, where: 0 = no pain and 10 = the worst pain imaginable. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use, where: 0 = no difficulty and 10 = so difficult it requires help.
  Scoring instructions: The scores from both dimensions are averaged to derive a total score.
Time Frame: Baseline and 12 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 48 | 87
units on a scale | -17.871 (2.477) | -10.554 (1.830)
Statistical Analysis 1: Comparison: Control vs Investigational; The null hypothesis (Ho) is that the effect of the two treatment groups at 12 weeks is equal and the corresponding alternative (Ha) is that the effect of the two treatment groups at 6 months is unequal; Test type: Superiority or Other; p = 0.018, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = 7.317, 95% CI 2-sided [1.249 to 13.386]

11. Secondary Outcome: Shoulder Pain and Disability Index (SPADI) Total Disability Score Change From Baseline and 12 Weeks (As Treated)
Description: as for outcome 10
Time Frame: Baseline and 12 weeks
Population: The As Treated analysis population included all subjects that received treatment and had outcome data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 68 | 129
units on a scale | -11.828 (2.132) | -9.467 (1.531)
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.369, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = 2.361, 95% CI 2-sided [-2.801 to 7.522]

12. Primary Outcome: Visual Analog Scale (VAS) Pain Score (As Treated)
Description: as for outcome 1
Time Frame: 6 Months
Population: The As Treated analysis population included all subjects that received treatment and had outcome data.
Measure: Least Squares Mean (Standard Error); unit: mm on a 100 mm VAS scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 64 | 132
mm on a 100 mm VAS scale | 33.196 (2.777) | 30.406 (1.926)
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.410, Mixed Models Repeated Measures ANCOVA — The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = -2.790, 95% CI 2-sided [-9.441 to 3.861]

13. Secondary Outcome: Shoulder Pain and Disability Index (SPADI) Total Disability Score Change From Baseline and 6 Months (Per Protocol)
Description: as for outcome 10
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 55 | 102
units on a scale | -16.109 (2.390) | -13.492 (1.752)
Statistical Analysis 1: Comparison: Control vs Investigational; The null hypothesis (Ho) is that the effect of the two treatment groups at 6 months is equal and the corresponding alternative (Ha) is that the effect of the two treatment groups at 6 months is unequal; Test type: Superiority or Other; p = 0.379, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = 2.617, 95% CI 2-sided [-3.226 to 8.460]

14. Secondary Outcome: Shoulder Pain and Disability Index (SPADI) Total Disability Score Change From Baseline and 6 Months (As Treated)
Description: as for outcome 10
Time Frame: Baseline and 6 months
Population: The As Treated analysis population included all subjects that received treatment and had outcome data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 63 | 127
units on a scale | -10.314 (2.179) | -12.522 (1.539)
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.409, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = -2.208, 95% CI 2-sided [-7.455 to 3.039]

15. Secondary Outcome: 12-Item Short Form Survey (SF-12) Physical Score Change From Baseline and 12 Weeks (Per Protocol)
Description: The difference in 12-Item Short Form Survey (SF-12) Physical score calculated as visit score - baseline score.
  The SF-12 is a generic measure and does not target a specific age or disease group. It has been developed to provide a shorter, yet valid alternative to the SF-36, which has been seen by many health researchers as too long to administer to studies with large samples. The SF-12 is weighted and summed to provide easily interpretable scales for physical and mental health.
  Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Baseline and 12 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 48 | 90
units on a scale | 3.607 (1.050) | 2.050 (0.771)
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.232, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = -1.558, 95% CI 2-sided [-4.119 to 1.003]

16. Secondary Outcome: 12-Item Short Form Survey (SF-12) Physical Score Change From Baseline and 12 Weeks (As Treated)
Description: as for outcome 15
Time Frame: Baseline and 12 weeks
Population: The As Treated analysis population included all subjects that received treatment and had outcome data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 67 | 133
units on a scale | 2.179 (0.877) | 1.950 (0.624)
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.832, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = -0.228, 95% CI 2-sided [-2.343 to 1.887]

17. Secondary Outcome: 12-Item Short Form Survey (SF-12) Physical Score Change From Baseline and 6 Months (Per Protocol)
Description: as for outcome 15
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 55 | 102
units on a scale | 2.763 (1.009) | 2.831 (0.743)
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.957, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = 0.068, 95% CI 2-sided [-2.396 to 2.532]

18. Secondary Outcome: 12-Item Short Form Survey (SF-12) Physical Score Change From Baseline and 6 Months (As Treated)
Description: as for outcome 15
Time Frame: Baseline and 6 months
Population: The As Treated analysis population included all subjects that received treatment and had outcome data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 63 | 126
units on a scale | 1.559 (0.896) | 2.779 (0.635)
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.267, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = 1.220, 95% CI 2-sided [-0.937 to 3.378]

19. Secondary Outcome: 12-Item Short Form Survey (SF-12) Mental Score Change From Baseline and 12 Weeks (Per Protocol)
Description: The difference in 12-Item Short Form Survey (SF-12) Mental score calculated as visit score - baseline score.
  The SF-12 is a generic measure and does not target a specific age or disease group. It has been developed to provide a shorter, yet valid alternative to the SF-36, which has been seen by many health researchers as too long to administer to studies with large samples. The SF-12 is weighted and summed to provide easily interpretable scales for physical and mental health.
  Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Baseline and 12 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 48 | 90
units on a scale | -0.130 (0.991) | 1.060 (0.726)
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.333, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = 1.190, 95% CI 2-sided [-1.225 to 3.604]

20. Secondary Outcome: 12-Item Short Form Survey (SF-12) Mental Score Change From Baseline and 12 Weeks (As Treated)
Description: as for outcome 19
Time Frame: Baseline and 12 weeks
Population: The As Treated analysis population included all subjects that received treatment and had outcome data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 67 | 133
units on a scale | 0.167 (0.875) | 0.938 (0.623)
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.473, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = 0.771, 95% CI 2-sided [-1.339 to 2.881]

21. Secondary Outcome: 12-Item Short Form Survey (SF-12) Mental Score Change From Baseline and 6 Months (Per Protocol)
Description: as for outcome 19
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 55 | 102
units on a scale | 0.397 (0.941) | 0.379 (0.692)
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.988, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = -0.018, 95% CI 2-sided [-2.314 to 2.278]

22. Secondary Outcome: 12-Item Short Form Survey (SF-12) Mental Score Change From Baseline and 6 Months (As Treated)
Description: as for outcome 19
Time Frame: Baseline and 6 months
Population: The As Treated analysis population included all subjects that received treatment and had outcome data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Control | Investigational
Number analyzed (Participants) | 63 | 126
units on a scale | 0.330 (0.897) | 0.798 (0.636)
Statistical Analysis 1: Comparison: Control vs Investigational; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.671, Mixed Models Repeated Measures ANCOVA — The p-value was not adjusted for multiple comparisons. The a priori threshold for significance was a two-sided p <0.05; The analysis included baseline score as a covariate. Site was dropped from the model due to statistical insignificance; Adjusted Mean Difference = 0.467, 95% CI 2-sided [-1.692 to 2.627]

ADVERSE EVENTS:
Time Frame: The first subject was randomized and treated in January, 2007. The last subject completed the study in August, 2010. Total timeframe: 3 years, 7 months
Description: All subjects that received study treatment are included in the safety population.
Groups:
- Control: Each subject received a one-time injection containing 6 mL of anesthetic (Marcaine)and 2 mL of corticosteroid (Celestone).
Arm/Group | Control | Investigational
Serious Adverse Events (participants affected / at risk) | 3/87 | 10/183
Other Adverse Events (participants affected / at risk) | 6/87 | 19/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=87) | Investigational (N=183)
Chest Pain - Cardiac Cath to Rule Out Cad (Cardiac disorders) | 0 (0) | 1 (1) — Angina pectoris
Knee Pain Both Knees (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Arthralgia
Shoulder Pain (Index Shoulder) Right Shoulder (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) — Musculoskeletal pain
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Breast Cancer Female
Patient has cancer, did not specify to PI where cancer is, never returned, lost to follow-up (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Neoplasm malignant
Total Shoulder Arthroplasty Plus Bone Graft Glenoid Scapular Right Shoulder (Surgical and medical procedures) | 0 (0) | 2 (2) — Shoulder Arthroplasty
Left Shoulder Pain Non-Study Shoulder - Surgery 6/10/09 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Musculoskeletal pain
Quadruple Bypass 5/6/09 (Surgical and medical procedures) | 1 (1) | 0 (0) — Coronary artery bypass
Iliopsoas Abscess (Infections and infestations) | 1 (1) | 0 (0) — Abscess
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Back pain
Open Heart Surgery After Aortic Valve Disease (Cardiac disorders) | 0 (0) | 1 (1) — Aortic valve disease
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=87) | Investigational (N=183)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 19 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days